CLINICAL TRIAL: NCT04640766
Title: Feasibility Open Label Study Evaluating the Use of Process-instructed Self Neuro-Modulation (PRISM) for Attention Deficit/ Hyperactivity Disorder - Adults
Brief Title: Process-instructed Self Neuro-Modulation (PRISM) for Attention Deficit/ Hyperactivity Disorder - Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-01086
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Attention Deficit Hyper Activity
Keywords: PRISM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants with ADHD (Experimental)
  Interventions: Device: PRISM

INTERVENTIONS:
Device: PRISM — The study will include 12 EEG-NF sessions, administered twice per week for a duration of 6 "active" weeks in total. Twice weekly sessions will be held on no-consecutive days. Each session will last approximately 30 minutes.
  Other Names: EEG-based neurofeedback (EEG-NF) device

SUMMARY:
This is a single-arm, open-label feasibility study. Participants will be assigned and will undergo a novel neurofeedback intervention, targeting down-regulation of deep limbic structures, specifically the amygdalae. Participants will complete 12 neurofeedback sessions delivered twice weekly over 6 consecutive weeks. The intervention will be delivered via the PRISM platform.

DETAILED DESCRIPTION:
The objectives include: 1)Training the NYU team on the electric finger print electroencephalography neurofeedback (EFP-EEG-NF) technology and provide them with hands-on experience; 2) Assessing participants' ability to learn the feedback paradigm (i.e. control the EFP-EEG-NF signal; time to achieve learning; assess learning curves); 3) Exploring preliminary results assessing target symptoms (e.g. AISRS and BRIEF-A).

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-60 years, inclusive at the time of consent
* Able to provide signed informed consent
* Any gender
* Subjects with a current primary DSM-5 diagnosis of ADHD (including predominantly inattentive presentation, hyperactive presentation, or combined presentations) as confirmed by the ACDS Version 1.2.
* Subjects who are not receiving any pharmacological treatment for ADHD must have an AISRS score of ≥ 28 at screening. Subjects who are receiving pharmacological treatment for ADHD at screening must have a minimum AISRS score of ≥ 22 at screening
* Not requiring treatment for any comorbid psychiatric condition for at least 2 months
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing
* No intention of changing medication or psychotherapy for the duration of the study at the time of recruitment

Exclusion Criteria:

* Concurrent substance abuse and/or history of substance use within 6 months
* Use of any prescribed benzodiazepine
* Lifetime bipolar disorder, psychotic disorder, autism, intellectual disability. Comorbid mood and anxiety disorders determined by the MINI will be permitted if they are not the primary focus of clinical attention
* Active suicidality within past year, or history of suicide attempt in past 2 years
* Any history of severe past drug dependence determined by the MINI (i.e., a focus of clinical attention or a cause of substantial social or occupational difficulty)
* Any unstable medical or neurological condition
* Any history of brain surgery, of penetrating, neurovascular, infectious, or other major brain injury, of epilepsy, or of other major neurological abnormality (including a history of traumatic brain injury [TBI] with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days)
* Any psychotropic medication
* Recent initiation (within the past 3 months) of cognitive-behavioral therapy or any evidence-based PTSD psychotherapy (Cognitive Processing Therapy [CPT], Prolonged Exposure [PE], Eye Movement Desensitization and Reprocessing [EMDR]); continuation of established maintenance supportive therapy will be permitted
* Significant hearing loss or severe sensory impairment
* Enrollment in another research study testing an experimental, clinical, or behavioral intervention intended to affect symptoms initiated within the last 2 months, or intended enrollment within the next 2.5 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Lenard.Adler@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants were enrolled; 9 of these participants failed screening. 9 participants started treatment.
Period: Overall Study
Arm/Group | Participants With ADHD
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawn for inconsistency with visits and change in current medication | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises individuals who began treatment in the study (n = 9).
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Score on Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: ADHD symptoms will also be measured using the Adult ADHD Investigator Symptom Rating Scale (AISRS). Items are scored as follows: 0 (none), 1 (mild), 2 (moderate), 3 (severe). The maximum total score for the scale is 54 points, with 27 points for each subscale. The total score is the sum of the inattentive and hyperactive-impulsive subscales. The higher the score, the more severe the symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
score on a scale | 35 (5.5)

2. Primary Outcome: Score on Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: as for outcome 1
Time Frame: Week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
score on a scale | 11.3 (6.9)

3. Primary Outcome: Score on Attention-Deficit/Hyperactivity Disorder Self-Report Screening Scale for DSM-5-Expanded (DSM-5 ASRS Expanded)
Description: The DSM-5 ASRS Expanded consists of 18 questions. Each question is scored in the range 0-4, for a total range of score of 0-72. The higher the score, the more difficulty the participant is experiencing handling ADHD.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
score on a scale | 47.1 (3.3)

4. Primary Outcome: Score on Attention-Deficit/Hyperactivity Disorder Self-Report Screening Scale for DSM-5-Expanded (DSM-5 ASRS Expanded)
Description: as for outcome 3
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
score on a scale | 32.4 (6.4)

5. Primary Outcome: Score on Behavioral Rating Inventory of Executive Function- Adult Version (BRIEF-A) Self-report
Description: Severity of executive function will be assessed via the Behavioral Rating Inventory of Executive Function- Adult version (BRIEF-A) self-report. All 75 items are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The total range of score is 0-150; higher scores indicate poor executive function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
score on a scale | 75.6 (7.6)

6. Primary Outcome: Score on Behavioral Rating Inventory of Executive Function- Adult Version (BRIEF-A) Self-report
Description: as for outcome 5
Time Frame: Week 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With ADHD
Number analyzed (Participants) | 9
score on a scale | 56.9 (9.6)

ADVERSE EVENTS:
Time Frame: 11 Weeks
Description: PI monitored for adverse events at every follow-up visit.
Arm/Group | Participants With ADHD
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With ADHD (N=9)
Insomnia + Vivid Dreams (Psychiatric disorders) | 1
Soreness in Jaw (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Gastrointestinal discomfort (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04640766/Prot_SAP_000.pdf